CLINICAL TRIAL: NCT00111137
Title: A Randomized, Open Label Study to Assess Time to Hemoglobin Response of a Front Load Dosing Regimen for Darbepoetin Alfa Compared to a Weekly Dose Regimen for Recombinant Human Erythropoietin in Patients With Non-Myeloid Malignancies Receiving Chemotherapy
Brief Title: Treatment for Patients With Non-Myeloid Malignancies Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20020139
Record Dates: First submitted 2005-05-17; First posted 2005-05-18 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2008-02

CONDITIONS: Cancer; Non-Myeloid Malignancies
Keywords: darbepoetin alfa; anemia; Amgen; Chemotherapy
MeSH Terms: conditions — Neoplasms; Anemia | interventions — Darbepoetin alfa

ARMS (2):
- rHuEPO (Active Comparator)
  Interventions: Drug: rHuEPO
- Darbepoetin alfa (Experimental)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: rHuEPO — rHuEPO 40,000U QW for 4 weeks. Dose will be increased to 60,000U/week at week 5 if inadequate response through week 12.
  Arms: rHuEPO
Drug: Darbepoetin alfa — 4.5 mcg/kg QW for 4 weeks then Q3W starting at week 5 through week 11.
  Arms: Darbepoetin alfa

SUMMARY:
The purpose of this study is to compare the time to hematopoietic response (hemoglobin correction to 12 g/dL or a greater than or equal to 2 g/dL increase from baseline) for subjects randomized to receive darbepoetin alfa with a front load dosing regimen to those receiving recombinant human erythropoietin (rHuEPO) with a weekly dose regimen during the 12-week comparative treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with non-myeloid malignancies planning to receive cyclic chemotherapy for 8 additional weeks or more
* Anemia (hemoglobin [hgb] greater than or equal to 9.0g/dL and less than or equal to 11.0 g/dL) related to cancer and chemotherapy
* Karnofsky performance status of greater than or equal to 50%
* Serum bilirubin less than or equal to 2.5 times the upper limit of normal range and serum creatinine concentration of less than or equal to 2.0 mg/dL

Exclusion Criteria:

* Acute myelogenous leukemia (AML), chronic myelogenous leukemia (CML), or myelodysplastic syndromes
* Hematologic disorder previously associated with anemia
* Active bleeding
* Iron deficiency
* Received erythropoietic therapy within 14 days prior to randomization
* Unstable cardiac disease
* Known positive human immunodeficiency virus antibody or hepatitis B surface antigen
* Known positive antibody response to any erythropoietic agent
* Currently enrolled in, or has not yet completed at least 30 days since ending other investigational device or drug trial or is receiving investigational agent(s) not approved for any indication
* Pregnant or breast feeding
* Red blood cell (RBC) transfusion within 4 weeks of screening
* Known hypersensitivity to any recombinant mammalian-derived product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2003-02; Primary Completion 2003-11 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Time to hematopoietic response during the comparative treatment period | during the comparative treatment period

SECONDARY OUTCOMES:
Exploratory analyses for other patient reported outcome scales collected during the study (FACT-Anemia, BSI, EQ-5D, and Patient Satisfaction Questionnaire for Injectable Anemia Treatment) | during the study
Incidence, if any, of neutralizing antibody formation to study drug | throughout study
Difference between the average hemoglobin after the first month of treatment compared to the baseline hemoglobin | baseline to first month of treatment
Time to 2 g/dL increase in hemoglobin during the comparative treatment period | during the comparative treatment period
Change in FACT-Fatigue scale score over time during the comparative treatment period | during the comparative treatment period
Overall incidence of adverse events, serious adverse events and related adverse events as measured throughout study | throughout study
Slope of change in hemoglobin after the first month of treatment | baseline to first month of treatment
Red blood cell usage during the treatment period and other changes in hemoglobin during the comparative treatment period | during the comparative treatment period
Changes in hemoglobin during the maintenance period | during the maintenance period

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com